CLINICAL TRIAL: NCT05627076
Title: Comparison of PSP Values Measured With Venous Whole Blood and Those Measured With Arterial Whole Blood.
Brief Title: Analytical Validation of the abioSCOPE Device With the IVD CAPSULE PSP Test: Comparison of PSP Values Measured With Venous Whole Blood and Those Measured With Arterial Whole Blood.
Status: Completed | Type: Observational
Sponsor: Abionic SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-PSP-006
Record Dates: First submitted 2022-11-10; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Sepsis; Sepsis Bacterial
Keywords: Abionic; Pancreatic Stone Protein; Point-of-care device; Immunoassay; IVD
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Blood Sampling — Blood samples will be collected for the PSP measurement using the abioSCOPE.

SUMMARY:
Abionic has developed a targeted, rapid test for pancreatic stone protein (PSP) in human K2-EDTA venous whole blood using the abioSCOPE instrument.

Currently no PSP study comparaison has been done between venous and arterial whole blood. Abionic would like to confirm the equivalence of the PSP between venous whole blood and arterial whole blood.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated written informed consent by patient or close / family / trusted person prior to any mandatory study-specific procedures, sample collection, or analysis;
2. Male or female, 18 years of age or older;
3. Patient admitted to hospital
4. Need for venous and arterial blood samples as part of standard of care
5. Covered by a social security scheme.

Exclusion Criteria:

1. Subject suffering from a hematological pathology (coagulation disorder, severe anemia) that could interfere with the blood draw procedure;
2. Subject under juridical protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted at the hospital
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Primary assessment | through study completion, an average of 1.5 months
  Pairwise comparability of test results when performed with K2-EDTA anticoagulated venous whole blood or K2-EDTA anticoagulated arterial whole blood, represented as percent recovery of arterial whole blood compared to venous whole blood, as well as scatter plots with Weighted Deming and Passing Bablok Regression, and bias plots.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Limoges, Réanimation Polyvalente, Limoges, France

IPD SHARING:
Plan to Share IPD: No